CLINICAL TRIAL: NCT02496936
Title: Acute Effects of Fats on Satiety and Energy Needs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: GFHNRC508
Record Dates: First submitted 2015-07-07; First posted 2015-07-14 (Estimated); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Obesity
Keywords: Energy Expenditure; Appetite; Satiety
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Saturated Fat (SFA) (Experimental): 30 grams saturated fat in the form of heavy whipping cream will be provided to subject in a smoothie drink
  Interventions: Other: SFA
- Monounsaturated Fat (MUFA) (Experimental): 30 grams monounsaturated fat in the form of high oleic canola oil will be provided to subject in a smoothie drink
  Interventions: Other: MUFA
- Polyunsaturated Fat Linoleic (PUFA-LA) (Experimental): 30 grams polyunsaturated fat in the form of high linoleic sunflower oil will be provided to subject in a smoothie drink
  Interventions: Other: PUFA-LA
- Polyunsaturated Fat Alpha-Linolenic (ALA) (Experimental): 30 grams polyunsaturated fat in the form of flaxseed oil will be provided to subject in a smoothie drink
  Interventions: Other: ALA
- Polyunsaturated Fat Long Chain Omega-3 (LCn3) (Experimental): 30 grams polyunsaturated fat in the form of fish oil (Coromega Omega3 Squeeze) will be provided to subject in a smoothie drink
  Interventions: Other: LCn3

INTERVENTIONS:
Other: SFA — High saturated fatty acid/SFA oil source
  Arms: Saturated Fat (SFA)
Other: MUFA — High monounsaturated fatty acid/MUFA oil source
  Arms: Monounsaturated Fat (MUFA)
Other: PUFA-LA — High polyunsaturated fatty acid (linoleic)/PUFA-LA oil source
  Arms: Polyunsaturated Fat Linoleic (PUFA-LA)
Other: ALA — High polyunsaturated fatty acid (alpha-linolenic)/ALA oil source
  Arms: Polyunsaturated Fat Alpha-Linolenic (ALA)
Other: LCn3 — High polyunsaturated fatty acid (omega-3)/LCn3 oil source
  Arms: Polyunsaturated Fat Long Chain Omega-3 (LCn3)

SUMMARY:
The purpose of this study is to assess the acute effect of dietary fat on satiety and energy metabolism.

DETAILED DESCRIPTION:
The influences of specific dietary fat sources on satiety, appetite and energy utilization remains unclear; evidence is lacking on whether responses vary according to acute intake. The researchers will use a controlled setting to determine whether the source of dietary fat is related to perceived satiety, satiety hormone responses, and energy expenditure by conducting experiments to evaluate short term (acute) effects.

ELIGIBILITY:
Inclusion Criteria:

* body mass index between 18.0-34.9 kg/m2
* free of major diagnosed, untreated medical conditions
* controlled hypertension
* non-smoking or use of other tobacco products, including e-cigarettes
* not taking steroid-based medications
* not planning to or currently attempting to gain or lose weight
* willing to comply with study demands
* use of oral contraceptives
* low intake of long chain omega 3 fatty acids

Exclusion Criteria:

* diagnosed eating disorders
* diabetes (blood sugar ≥ 126 mg/dl)
* hypertension (systolic ≥ 160 mmHg or diastolic > 100 mmHg)
* diagnosed cardiovascular, pulmonary, skeletal and metabolic disease
* currently pregnant or planning to become pregnant, or lactating
* taking medications known to affect appetite, blood lipids, body composition, body weight, or food intake (appetite control drugs, steroids, antidepressants)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Acute effect of fat intake on energy expenditure as determined by metabolic rate | Incremental Area Under the Curve (iAUC) of metabolic rate from 0 to 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Picklo, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Grand Forks Human Nutrition Research Center Current Nutrition Studies — https://www.ars.usda.gov/plains-area/gfnd/gfhnrc/docs/nutrition-studies/nutrition-studies/

DOCUMENTS (1):
  • Informed Consent Form (2019-09-06): https://cdn.clinicaltrials.gov/large-docs/36/NCT02496936/ICF_000.pdf